CLINICAL TRIAL: NCT02450513
Title: Adalimumab Trough Concentrations in Crohn's Disease: A Pilot Pharmacokinetic Study
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S53297
Record Dates: First submitted 2015-05-12; First posted 2015-05-21 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Crohn's Disease
Keywords: adalimumab; anti-TNF; pharmacokinetics; trough level; immunogenicity
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Single-group study: Subjects with active refractory Crohn's disease naïve to TNF antagonists starting adalimumab therapy.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — 160 mg at week 0, 80 mg at week 2 and 40 mg every two weeks onwards
  Other Names: Humira

SUMMARY:
Observational pharmacokinetics study of adalimumab in patients with active refractory Crohn's disease who are naïve to TNF antagonist therapy.

DETAILED DESCRIPTION:
Adalimumab (ADM), a fully human tumor necrosis factor (TNF) antagonist, is effective for treating patients with Crohn's disease (CD). A correlation between concentration and effect was observed at distinct time points.

The aim was to evaluate the correlation of early longitudinal measurements of ADM with different biological markers for disease activity and induction and maintenance of clinical remission.

This is a prospective two-center open-label observational study in anti-TNF naïve patients with moderate to severe CD induced with ADM 160/80 mg at week 0 and 2 and 40 mg every 2 weeks in monotherapy. All patients should be in need for TNF antagonist therapy and should fulfill standard reimbursement criteria (Belgium). Serum samples were taken pre and post first injection and at weeks 1, 2, 3, 4, 12, 26 and 52. Following parameters were determined: C-reactive protein, albumin, TNF, ADM, antibodies to ADM, hemoglobin, platelet count and leukocyte count. Clinical response and remission was evaluated using the Harvey-Bradshaw index.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of Crohn's disease, fulfilling the criteria for reimbursement (Belgium).
* Patients with active disease defined as a Harvey-Bradshaw index >4 and/or a C-reactive protein concentration >5 mg/l.
* Informed consent.

Exclusion Criteria:

* Patients with ulcerative colitis.
* Patients treated in placebo controlled trials.
* Patients unwilling to participate or withdrawing informed consent for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are naïve to TNF antagonist treatment and who will be started on adalimumab for treatment of active refractory Crohn's disease. All patients should be in need for TNF antagonist therapy and should fulfill standard reimbursement criteria (Belgium).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-03; Primary Completion 2016-05-25 (Actual); Study Completion 2016-05-25 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in clinical remission | week 12
  As defined by a Harvey-Bradshaw index ≤4

CONTACTS AND LOCATIONS:
Overall Officials: Filip Baert, MD, Principal Investigator — Filip.Baert@azdelta.be
Locations (2):
- Belgium (2):
  - University Hospitals Leuven, Leuven
  - AZ Delta, Roeselare

REFERENCES:
- [Derived] Vande Casteele N, Baert F, Bian S, Dreesen E, Compernolle G, Van Assche G, Ferrante M, Vermeire S, Gils A. Subcutaneous Absorption Contributes to Observed Interindividual Variability in Adalimumab Serum Concentrations in Crohn's Disease: A Prospective Multicentre Study. J Crohns Colitis. 2019 Sep 27;13(10):1248-1256. doi: 10.1093/ecco-jcc/jjz050. PMID 30820530